CLINICAL TRIAL: NCT06147310
Title: Effect of Albumin Gel-platelet-rich Fibrin (Alb-PRF) and Advanced Platelet-rich Fibrin (A-PRF) in Alveolar Ridge Preservation in Diabetes Patients - A Randomized Controlled Clinical Trial
Brief Title: Effect Alb-PRF & A-PRF in Alveolar Ridge Preservation in Diabetes Patients - A RCCT
Acronym: AlbPRFARP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Melissa Fok, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L2023_01
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Tooth Extraction Status Nos
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective, parallel group, randomized-controlled, single-blinded, superiority clinical study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participlant will be masked Care provider and investigator could not be masked due to the intrinsic nature of the intervention, however the allocation will be concealed until the extraction of teeth is completed.
  Outcome assessor will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Alveolar ridge preservation with Alb-PRF + A-PRF after extraction
  Interventions: Procedure: Study Group
- Control Group (Placebo Comparator): Spontaneous healing after extraction
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: Study Group — The tooth will be extracted automatically, tooth sectioning will be performed if necessary for multi-rooted teeth to minimize trauma. Alveolar ridge preservation with blood platelet concentrate: heat-treated albumin (Alb-PRF) and advanced platelet-rich fibrin. The experimental site will be filled with A-PRF plugs/membranes until level flushed with the level of bone. An additional Alb-PRF membrane will be tucked and inserted below the buccal and oral flap. Surgical flaps will not be raised. Soft tissue will be tunnelled and undermined for insertion of the Alb-PRF membrane. The extraction site and membranes will be stabilized by cross-mattress sutures and allowed for secondary intention healing.
  Other Names: Albumin-platelet rich fibrin, Advanced platelet rich fibrin
  Arms: Study Group
Procedure: Control Group — The tooth will be extracted automatically, tooth sectioning will be performed if necessary for multi-rooted teeth to minimize trauma. Cross mattress suture will be applied and site allowed to heal naturally.
  Arms: Control Group

SUMMARY:
This study aim to investigate the effect of albumin gel- and platelet- rich fibrin(Alb-PRF) combined with advanced platelet-rich fibrin (A-PRF) on alveolar ridge preservation by comparing alveolar ridge morphometric changes (hard and soft tissue), prospects and treatment complexity for placement of prosthetically guided dental implant, early oral wound healing outcomes evaluated by the Inflammatory Proliferative Remodeling Scale, and patient reported outcome measures, in Type I/II Diabetes Mellitus patient, versus spontaneous healing

DETAILED DESCRIPTION:
Diabetes is a well-established risk factor for oral diseases that often lead to extractions and tooth loss in the population, while diabetic patients also have increased susceptibility to wound infections.

Albumin gel-platelet-rich fibrin (Alb-PRF) and advanced platelet-rich fibrin (A-PRF) are third-generation of platelet concentrates derived from a donor's blood by following a simple centrifugation protocol, heat treatment of platelet-poor plasma, and mixing of liquid-PRF from the same preparation.

This study proposes a novel alveolar ridge preservation technique based on the application of A-PRF inside the extraction socket to sustain the release of growth factors during the early wound healing phase, together with periosteum inhibition by overlaying an Alb-PRF membrane with slow biodegradation and space maintenance properties over the bone to reduce post-extraction alveolar ridge resorption.

ELIGIBILITY:
i. At least 18 years old with established TIIDM diagnosis for more than 0.5 years, fasting blood glucose ≥7.0 mmol/L or 2 h plasma glucose ≥11.1 mmol/L, maximum HbA1c levels under 8.0%.

ii. Non-smoker, diagnosed with generalized periodontitis stage III or IV. iii. Need for extraction of teeth, on opposing arches or opposing sides, with or without other concurrent indications for extractions: orthodontics, periodontitis, caries, fracture, root resorption, unrestorable root fragments.

iv. At least one adjacent teeth/ implant is present at the site of extraction with a secure prognosis.

v. No periapical lesions with a diameter of more than 5 mm (radiographically determined.

vi. Extraction socket with a bone height of at least 7mm at 2 walls. vii. Reasonably aligned dental arches viii. Will consider implant to replace missing teeth ix. Willing and able to give informed consent.

Exclusion Criteria:

i. Patients with conditions or circumstances, in the opinion of the Investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance or unreliability.

ii. Pregnancy or intention to become pregnant at any point during the study duration.

iii. Smoker /alcoholic iv. Has platelet dysfunction/ thrombocytopenia/ blood dyscrasia v. On bisphosphonates or drugs that will significantly alter bone metabolism. vi. ASA III/IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Ridge horizontal width | Up to 20 weeks
  Ridge horizontal width changes (1mm, 3mm, 5mm apical to most coronal crest at buccal/oral) Method: CBCT

SECONDARY OUTCOMES:
Ridge height | Up to 20 weeks
  Ridge height changes (buccal and oral) Method: CBCT
Ridge volume and profile | Up to 20 weeks
  Changes in ridge volume and profilometric changes Method: Intraoral scan, CBCT
Keratinized tissue width changes | Up to 20 weeks
  Changes in keratinized tissue width Method: Periodontal probe with fixed landmarks
Cytokines and growth factors | Up to 56 days
  Changes in concentrations of cytokines and growth factors in wound fluid during early to mid-term wound healing events
Implant planning related outcome | Up to 20 weeks
  Ability to place prosthetically guided implant, need for additional augmentation
Histological assessment | Up to 24 weeks
  Bone volume to total tissue volume ratio and bone microstructure Method: Core biopsy with trephine at day of implant placement, micro CT and histomorphometric assessment
Patient-reported outcome measures | Up to 28 days
  Patient will be asked to record their pre-operative anxiety level, intraoperative pain level and pain levels at follow up visits on a visual analogue scale (0-10)
Inflammatory proliferative remodelling | Up to 28 days
  IPR score will be assessed by independent assessors with photos of wound site at different itme points

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Fok, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No